CLINICAL TRIAL: NCT03845205
Title: Alcohol Treatment Outcomes Following Early vs. Standard Liver Transplant for Severe Alcoholic Hepatitis (SAH)
Brief Title: Alcohol Treatment Outcomes Following Early vs. Standard Liver Transplant for SAH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00152700; P50AA027054 (NIH)
Record Dates: First submitted 2019-02-15; First posted 2019-02-19 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Alcohol Use Disorder; Alcoholic Hepatitis
Keywords: Alcohol treatment; Liver transplant; Motivational intervention; Cognitive-behavioral therapy
MeSH Terms: conditions — Alcoholism; Hepatitis, Alcoholic | interventions — Ethanol; Methods

STUDY DESIGN:
Intervention Model Description: Integrated AUD treatment (IAT) v Treatment as usual (TAU)
Who Masked: Outcomes Assessor
Masking Description: Research Coordinator is blinded to treatment assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated AUD Treatment (IAT) (Experimental): IAT will include computer-delivered CBI in the hospital, nurse-delivered clinical monitoring and treatment adherence counseling, and at-home participation in web-based, 7-session computerized cognitive-behavioral therapy (CBT4CBT), supplemented by tailored text messages. Alcohol pharmacotherapy will be added to behavioral treatments as needed.
  Interventions: Behavioral: Integrated AUD Treatment
- Treatment As Usual (No Intervention): All LT patients receive physician instructions to not drink alcohol. Consistent with current discharge procedures, AH patients are encouraged to engage in alcohol treatment services. Patients receive regular blood draws for monitoring of liver function, and regular phone calls for post-operative monitoring.

INTERVENTIONS:
Behavioral: Integrated AUD Treatment — IAT will include computer-delivered BI in the hospital, nurse-delivered alcohol monitoring counseling at each outpatient LT follow-up visit, and at-home participation in web-based, 7-session CBT4CBT, supplemented by tailored text messages.
  Other Names: Computerized brief alcohol intervention (CBI); CBT4CBT; Text Messaging
  Arms: Integrated AUD Treatment (IAT)

SUMMARY:
Given the severe consequences of alcohol relapse following liver transplantation for alcoholic hepatitis (AH-LT), it is critical to accurately identify alcohol use and implement alcohol interventions early in the post-transplant period to optimize patient outcomes. The proposed randomized clinical trial will examine the implementation and effects of integrated, person- and computer-delivered alcohol treatment compared to standard care on alcohol use (assessed by self-report and biomarker), mood, quality of life and survival following AH-LT. Predictors of 12-month post-transplant alcohol outcomes will be explored to allow future improved tailoring and targeting of these treatments.

DETAILED DESCRIPTION:
In the United States, alcoholic liver disease (ALD) is the second most common indication for liver transplant (LT). Traditionally, ALD patients have been required to complete a six-month mandatory period of alcohol abstinence before LT. More recently early LT for severe alcoholic hepatitis is being performed without any pre-transplant alcohol treatment because of the high medical acuity and mortality associated with this disease. Importantly, the limited studies to-date demonstrate comparable survival among early (ELT) versus standard (SLT) transplant recipients. Return to alcohol use is a major concern for all LT recipients with ALD, with estimates of alcohol relapse ranging between 16 and 49%. Although most LT clinics have enforced pre-LT alcohol treatment, far less attention has been paid to post-LT services, despite the high risk and severe consequences of relapse during this period. Numerous evidence-based treatments are available for alcohol use disorder (AUD). In recent years, the investigators and others have developed web- and text-based versions of these empirically-supported interventions to expand the reach and replicability outside of formal alcohol clinic settings. Delivery of AUD interventions in non-traditional settings is feasible, acceptable to patients, and effective in reducing alcohol use. The investigators propose to implement and evaluate the effects of alcohol treatment integrated into routine post-LT care. All patients receive physician instructions to stop drinking and engage in alcohol services (treatment as usual: TAU). ELT (N=100) and SLT (N=100) patients will be randomized on a 2:1 basis to integrated AUD treatment (IAT) or TAU. IAT will include computer-delivered BI in the hospital, nurse-delivered alcohol monitoring counseling at each outpatient LT follow-up visit, and at-home participation in web-based, 7-session CBT4CBT, supplemented by tailored text messages. Also, because of the evidence that ALD patients significantly underreport drinking to LT providers, the investigators will compare post-LT alcohol relapse rates using a well-validated biomarker of recent drinking (PEth), patient self-report on a validated alcohol instrument, and patient report to LT provider. Finally, the investigators will identify predictors of post-LT alcohol use and treatment engagement for ELT and SLT patients. Key measures will include: alcohol use; engagement in alcohol treatment; retention in post-transplant follow-up care; mood and anxiety; and quality of life. Given the severe consequences of alcohol relapse among both ELT and SLT recipients, it is critical to accurately identify alcohol use and implement alcohol interventions early in the post-transplant period to optimize short- and long-term patient outcomes and ultimately tailor treatments for this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* English speaking

Exclusion Criteria:

* too medically/psychiatrically ill to participate
* not able to provide informed consent due to cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-11-20 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Treatment engagement as assessed by proportion of kept LT follow-up appointments | 1 year
  Proportion of kept/scheduled LT follow-up appointments
Alcohol relapse as assessed by time to first Phosphatidyl ethanol (PEth) level ≥ 8 ng/mL | 1 year
  Time to first Phosphatidyl ethanol (PEth) level ≥ 8 ng/mL (minimum detectable level)
Post-liver transplant survival as assessed by time to death | 1 year
  Time to death (in months)

SECONDARY OUTCOMES:
Alcohol relapse as assessed by Timeline Followback Interview | 1 year
  Any alcohol use reported on the Timeline Followback Interview

CONTACTS AND LOCATIONS:
Overall Officials: Mary E McCaul, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee BP, Chen PH, Haugen C, Hernaez R, Gurakar A, Philosophe B, Dagher N, Moore SA, Li Z, Cameron AM. Three-year Results of a Pilot Program in Early Liver Transplantation for Severe Alcoholic Hepatitis. Ann Surg. 2017 Jan;265(1):20-29. doi: 10.1097/SLA.0000000000001831. PMID 27280501
- [Background] Weeks SR, Sun Z, McCaul ME, Zhu H, Anders RA, Philosophe B, Ottmann SE, Garonzik Wang JM, Gurakar AO, Cameron AM. Liver Transplantation for Severe Alcoholic Hepatitis, Updated Lessons from the World's Largest Series. J Am Coll Surg. 2018 Apr;226(4):549-557. doi: 10.1016/j.jamcollsurg.2017.12.044. Epub 2018 Feb 2. PMID 29409981
- [Background] Fleming MF, Smith MJ, Oslakovic E, Lucey MR, Vue JX, Al-Saden P, Levitsky J. Phosphatidylethanol Detects Moderate-to-Heavy Alcohol Use in Liver Transplant Recipients. Alcohol Clin Exp Res. 2017 Apr;41(4):857-862. doi: 10.1111/acer.13353. Epub 2017 Mar 20. PMID 28196282
- [Background] Chander G, Hutton HE, Lau B, Xu X, McCaul ME. Brief Intervention Decreases Drinking Frequency in HIV-Infected, Heavy Drinking Women: Results of a Randomized Controlled Trial. J Acquir Immune Defic Syndr. 2015 Oct 1;70(2):137-45. doi: 10.1097/QAI.0000000000000679. PMID 25967270
- [Background] Kiluk BD, Devore KA, Buck MB, Nich C, Frankforter TL, LaPaglia DM, Yates BT, Gordon MA, Carroll KM. Randomized Trial of Computerized Cognitive Behavioral Therapy for Alcohol Use Disorders: Efficacy as a Virtual Stand-Alone and Treatment Add-On Compared with Standard Outpatient Treatment. Alcohol Clin Exp Res. 2016 Sep;40(9):1991-2000. doi: 10.1111/acer.13162. Epub 2016 Aug 4. PMID 27488212